CLINICAL TRIAL: NCT01340937
Title: A Phase III Randomized, Partially Double-Blind, Active-Comparator-Controlled, Lot-to-Lot Consistency Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V419 in Healthy Infants When Given at 2, 4, and 6 Months Concomitantly With Prevnar 13™ and RotaTeq ™
Brief Title: A Study of V419 Given Concomitantly With Prevnar 13™ and RotaTeq™ (V419-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V419-006
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Bacterial Infections; Virus Diseases
Keywords: Diphtheria; Tetanus; Whooping Cough (pertussis); Poliomyelitis; Hepatitis B infection; Haemophilus influenzae type b infection
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections | interventions — pentacel; 13-valent pneumococcal vaccine; RotaTeq

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- V419 Lot A (Experimental): V419 (Lot A) 0.5 mL intramuscular injection (IM) at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 month of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age
  Interventions: Biological: V419; Biological: PENTACEL™; Biological: Prevnar 13™; Biological: RotaTeq™
- V419 Lot B (Experimental): V419 (Lot B) 0.5 mL IM at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 month of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age
  Interventions: Biological: V419; Biological: PENTACEL™; Biological: Prevnar 13™; Biological: RotaTeq™
- V419 Lot C (Experimental): V419 (Lot C) 0.5 mL IM at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 month of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age
  Interventions: Biological: V419; Biological: PENTACEL™; Biological: Prevnar 13™; Biological: RotaTeq™
- Control (Active Comparator): Pentacel™ 0.5 mL IM at 2, 4, 6, and 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age; and Recombivax HB vaccine 0.5 mL IM at 2 and 6 months of age
  Interventions: Biological: PENTACEL™; Biological: Prevnar 13™; Biological: RotaTeq™; Biological: Recombivax HB vaccine

INTERVENTIONS:
Biological: V419 — V419 (Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus, Haemophilus b Conjugate [Meningococcal Outer Membrane Protein Complex], and Hepatitis B [Recombinant] Vaccine) (from one of three lots) 0.5 mL intramuscular injection at 2, 4, and 6 months of age.
  Arms: V419 Lot A; V419 Lot B; V419 Lot C
Biological: PENTACEL™ — PENTACEL™ 0.5 mL intramuscular injection at 15 months of age in the V419 groups and at 2, 4, 6, and 15 months of age in the control group
Biological: Prevnar 13™ — Prevnar 13™ 0.5 mL intramuscular injection at 2, 4, 6, and 15 months of age
Biological: RotaTeq™ — RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age
Biological: Recombivax HB vaccine — Recombivax HB vaccine 0.5 mL intramuscular injection at 2 and 6 months of age
  Arms: Control

SUMMARY:
This study will determine whether three manufacturing lots of V419 (PR5I) induce similar immune responses to all of the antigens contained in V419 when given concomitantly with Prevnar13™ and RotaTeq™.

DETAILED DESCRIPTION:
This study is partially Double-Blinded in that the participants' parents/guardians, investigator/study site personnel, and Sponsor's representatives will be blinded to the lot of V419 the participant is randomized to receive, but not to the participant's treatment group (V419 or control).

ELIGIBILITY:
Inclusion Criteria :

* Participant is a healthy infant
* Participant has received one dose of monovalent hepatitis B vaccine prior to 1 month of age

Exclusion Criteria :

* Participant has received more than one dose of monovalent hepatitis B vaccine or hepatitis B based combination vaccine prior to study entry
* Participant has been vaccinated with any acellular pertussis or whole cell pertussis based combination vaccines, haemophilus influenzae type b conjugate, poliovirus, pneumococcal conjugate or pneumococcal polysaccharide, rotavirus, measles, mumps, rubella, or varicella vaccines or any combination of the above
* Participant has had an illness with fever within 24 hours of study enrollment
* Participant was vaccinated with any non-study vaccine (i.e. inactivated, conjugated or live virus vaccine within 30 days prior to enrollment, except for inactivated influenza vaccine, which is permitted 15 days or more prior to enrollment
* Participant or his/her mother has hepatitis B surface antigen (HBsAg) seropositivity (by medical history)
* Participant has a history of haemophilus influenzae type B, hepatitis B, diphtheria, tetanus, pertussis, poliomyelitis, rotavirus, or pneumococcal infection

Ages: 46 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2808 (Actual)
Dates: Start 2011-05-10 (Actual); Primary Completion 2012-12-18 (Actual); Study Completion 2013-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Block SL, Klein NP, Sarpong K, Russell S, Fling J, Petrecz M, Flores S, Xu J, Liu G, Stek JE, Foglia G, Lee AW. Lot-to-lot Consistency, Safety, Tolerability and Immunogenicity of an Investigational Hexavalent Vaccine in US Infants. Pediatr Infect Dis J. 2017 Feb;36(2):202-208. doi: 10.1097/INF.0000000000001405. PMID 27846058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The infant series of vaccinations were those administered at 2, 4, and 6 months of age; the toddler vaccinations were those administered at 15 months of age. The Interim Period is the time between the last vaccination of the infant series and the time of administration of the toddler vaccination.
Groups:
- V419 Lot A: V419 (Lot A) 0.5 mL intramuscular injection (IM) at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age.
- V419 Lot B: V419 (Lot B) 0.5 mL intramuscular injection (IM) at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age.
- V419 Lot C: V419 (Lot C) 0.5 mL intramuscular injection (IM) at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age.
Period: Period 1: Infant Series
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Started | 800 | 797 | 809 | 402
Completed | 742 | 737 | 753 | 370
Not Completed | 58 | 60 | 56 | 32
Not completed — Other protocol criterion not met | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 4 | 0
Not completed — Death | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 20 | 14 | 12 | 13
Not completed — Physician Decision | 2 | 3 | 1 | 0
Not completed — Protocol Violation | 1 | 4 | 4 | 3
Not completed — Withdrawal by Subject | 33 | 32 | 30 | 15
Not completed — Randomized but not vaccinated | 0 | 5 | 2 | 1
Period: Period 2: Interim Period
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Started | 742 | 737 | 753 | 370
Completed | 675 | 658 | 669 | 329
Not Completed | 67 | 79 | 84 | 41
Not completed — Withdrawal by Subject | 28 | 23 | 17 | 12
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 29 | 48 | 53 | 23
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 5 | 3 | 6 | 3
Not completed — Technical problems | 4 | 4 | 6 | 3
Period: Period 3: Toddler Vaccinations
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Started | 675 | 658 | 669 | 329
Completed | 666 | 641 | 660 | 319
Not Completed | 9 | 17 | 9 | 10
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 1
Not completed — Lost to Follow-up | 6 | 14 | 7 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Technical problem | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | Total
Number analyzed (Participants) | 800 | 797 | 809 | 402 | 2808
Age, Continuous [Mean (Standard Deviation); unit: Days] | 64.6 (6.7) | 64.4 (6.2) | 64.7 (6.6) | 64.3 (6.6) | 64.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 377 | 366 | 380 | 215 | 1338
  Male | 423 | 431 | 429 | 187 | 1470

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration of Antibodies to Polyribosylribitol Phosphate Antigen
Description: Participant serum samples were collected for testing with a radioimmunoassay for antibodies to Haemophilus influenza type b capsular polysaccharide polyribosylribitol phosphate.
Time Frame: Postdose 3 (Month 7)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had an infant vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- V419 Lots A, B, and C Combined: V419 (Lot A, B, or C) 0.5 mL intramuscular injection (IM) at 2, 4, and 6 months of age; Pentacel™ 0.5 mL IM at 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age.
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 604 | 596 | 595 | 288 | 1795
µg/mL | 5.51 [4.88 to 6.21] | 6.10 [5.38 to 6.92] | 6.59 [5.80 to 7.47] | 3.76 [3.11 to 4.55] | 6.05 [5.63 to 6.50]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the Geometric Mean Concentration (GMC) ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.91, 95% CI 2-sided [0.77 to 1.08] — GMC ratio was adjusted for post- and prevaccination titer, vaccination group, and brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 0.86, 95% CI 2-sided [0.72 to 1.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 0.94, 95% CI 2-sided [0.79 to 1.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; GMC, GMC ratio, and p-value were adjusted for post- and prevaccination titer, vaccination group, and brand of birth dose of Hepatitis B vaccine; GMC Ratio (Combined/Control) = 1.63, 95% CI 2-sided [1.35 to 1.98]

2. Secondary Outcome: Percentage of Participants Responding to Polyribosylribitol Phosphate Antigen
Description: Participant serum samples were collected for testing with a radioimmunoassay for antibodies to Haemophilus influenza type b capsular polysaccharide polyribosylribitol phosphate. Response was evaluated for a titer >=0.15 µg/mL and >=1.0 µg/mL.
Time Frame: Postdose 3 (Month 7)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had a vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 604 | 596 | 595 | 288 | 1795
Percentage of participants
  Titer >=1 µg/mL | 86.75 [83.79 to 89.36] | 87.25 [84.30 to 89.82] | 88.40 [85.55 to 90.86] | 79.51 [74.39 to 84.02] | 87.47 [85.84 to 88.96]
  Titer >=0.15 µg/mL | 99.01 [97.85 to 99.63] | 98.32 [96.94 to 99.19] | 97.82 [96.29 to 98.83] | 96.18 [93.27 to 98.08] | 98.38 [97.69 to 98.92]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Equivalence for titer >=1 µg/mL; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = -0.48, 95% CI 2-sided [-4.31 to 3.35] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Equivalence for titer >=1 µg/mL; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = -1.62, 95% CI 2-sided [-5.38 to 2.12] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Equivalence for titer >=1 µg/mL; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = -1.16, 95% CI 2-sided [-4.89 to 2.58] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Non-inferiority for titer >=1 µg/mL; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 7.93, 95% CI 2-sided [3.38 to 13.17]
Statistical Analysis 5: Comparison: Control vs V419 Lots A, B, and C Combined; Non-inferiority for titer >=0.15 µg/mL; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 2.20, 95% CI 2-sided [0.39 to 5.12]

3. Primary Outcome: Geometric Mean Concentration of Antibodies to Hepatitis B Surface Antigen
Description: Participant serum samples were collected for testing with an enhanced chemiluminescence assay for antibodies to Hepatitis B Surface Antigen. The unit of measure is milli International Units/mL (mIU/mL).
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Number analyzed (Participants) | 588 | 599 | 580 | 286
mIU/mL | 1195.96 [1081.62 to 1322.39] | 1376.86 [1264.74 to 1498.92] | 1414.52 [1297.52 to 1542.06] | 609.08 [515.29 to 719.93]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.87, 95% CI 2-sided [0.76 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 0.85, 95% CI 2-sided [0.74 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 0.98, 95% CI 2-sided [0.86 to 1.11] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Geometric Mean Concentration of Antibodies to Diphtheria Toxin
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to diphtheria toxin. The unit of measure is International Units/mL (IU/mL).
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Number analyzed (Participants) | 622 | 625 | 618 | 301
IU/mL | 0.37 [0.34 to 0.40] | 0.36 [0.33 to 0.40] | 0.38 [0.34 to 0.41] | 0.40 [0.35 to 0.45]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.95, 95% CI 2-sided [0.84 to 1.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 0.97, 95% CI 2-sided [0.86 to 1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 1.02, 95% CI 2-sided [0.90 to 1.14] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Geometric Mean Concentration of Antibodies to Tetanus Toxin
Description: Participant serum samples were collected for testing with an Enzyme-linked Immunosorbent Assay (ELISA) for anti-tetanus antibodies.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Number analyzed (Participants) | 622 | 609 | 612 | 300
IU/mL | 1.59 [1.51 to 1.67] | 1.63 [1.55 to 1.71] | 1.55 [1.48 to 1.63] | 0.89 [0.81 to 0.97]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.97, 95% CI 2-sided [0.91 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 1.02, 95% CI 2-sided [0.95 to 1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 1.05, 95% CI 2-sided [0.98 to 1.13] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. The unit of measure is ELISA units/mL (EU/mL).
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 647 | 634 | 622 | 309 | 1903
EU/mL | 100.83 [95.98 to 105.91] | 96.82 [92.10 to 101.79] | 98.52 [93.84 to 103.43] | 82.45 [77.26 to 87.98] | 98.72 [95.96 to 101.57]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 1.03, 95% CI 2-sided [0.96 to 1.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 1.02, 95% CI 2-sided [0.95 to 1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 0.99, 95% CI 2-sided [0.92 to 1.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Secondary analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.20, 95% CI 2-sided [1.11 to 1.29]

7. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 644 | 631 | 628 | 312 | 1903
EU/mL | 43.98 [41.45 to 46.66] | 49.19 [46.52 to 52.02] | 56.93 [53.73 to 60.31] | 73.25 [67.94 to 78.97] | 49.70 [48.06 to 51.40]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.89, 95% CI 2-sided [0.83 to 0.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 0.78, 95% CI 2-sided [0.72 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 0.87, 95% CI 2-sided [0.81 to 0.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Secondary analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p = 0.419, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.67, 95% CI 2-sided [0.62 to 0.73]

8. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 632 | 616 | 611 | 303 | 1859
EU/mL | 51.30 [47.46 to 55.44] | 52.32 [47.85 to 57.21] | 54.78 [50.33 to 59.61] | 50.96 [45.38 to 57.21] | 52.76 [50.27 to 55.37]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.97, 95% CI 2-sided [0.87 to 1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 0.93, 95% CI 2-sided [0.83 to 1.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 0.96, 95% CI 2-sided [0.85 to 1.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Secondary analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.03, 95% CI 2-sided [0.90 to 1.17]

9. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 641 | 632 | 623 | 309 | 1896
EU/mL | 228.78 [213.87 to 244.73] | 286.74 [268.86 to 305.81] | 283.28 [264.52 to 303.36] | 175.65 [159.14 to 193.87] | 264.61 [254.54 to 275.07]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot B) = 0.78, 95% CI 2-sided [0.72 to 0.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot A/Lot C) = 0.80, 95% CI 2-sided [0.73 to 0.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMC ratio are within the margin 0.67 to 1.5; GMC Ratio (Lot B/Lot C) = 1.02, 95% CI 2-sided [0.93 to 1.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Secondary analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.51, 95% CI 2-sided [1.37 to 1.66]

10. Primary Outcome: Geometric Mean Titer for Antibodies to Poliovirus Type 1
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 1. The unit of measure is titer (reciprocal of highest dilution with neutralizing activity).
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Number analyzed (Participants) | 630 | 632 | 628 | 307
Titer | 579.77 [533.82 to 629.68] | 684.68 [628.40 to 746.01] | 666.18 [612.30 to 724.79] | 269.95 [232.21 to 313.83]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the Geometric Mean Titer (GMT) ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot A/Lot B) = 0.86, 95% CI 2-sided [0.76 to 0.96] — GMT ratio was adjusted for post- and prevaccination titer, vaccination group, and brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot A/Lot C) = 0.88, 95% CI 2-sided [0.79 to 0.99] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot B/Lot C) = 1.03, 95% CI 2-sided [0.92 to 1.15] — [estimate comment as in outcome 10, analysis 1]

11. Primary Outcome: Geometric Mean Titer for Antibodies to Poliovirus Type 2
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 2.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Number analyzed (Participants) | 630 | 632 | 633 | 307
Titer | 1212.40 [1116.40 to 1316.65] | 1276.56 [1172.86 to 1389.43] | 1359.78 [1248.13 to 1481.42] | 846.14 [751.81 to 952.30]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot A/Lot B) = 0.94, 95% CI 2-sided [0.84 to 1.05] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot A/Lot C) = 0.91, 95% CI 2-sided [0.82 to 1.02] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot B/Lot C) = 0.98, 95% CI 2-sided [0.87 to 1.09] — [estimate comment as in outcome 10, analysis 1]

12. Primary Outcome: Geometric Mean Titer for Antibodies to Poliovirus Type 3
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 3.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control
Number analyzed (Participants) | 624 | 625 | 625 | 304
Titer | 901.70 [819.52 to 992.12] | 851.34 [772.96 to 937.66] | 825.31 [746.52 to 912.42] | 784.24 [682.28 to 901.44]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot A/Lot B) = 1.06, 95% CI 2-sided [0.92 to 1.22] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot A/Lot C) = 1.09, 95% CI 2-sided [0.95 to 1.26] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% confidence intervals of the GMT ratio are within the margin 0.67 to 1.5; GMT Ratio (Lot B/Lot C) = 1.03, 95% CI 2-sided [0.90 to 1.19] — [estimate comment as in outcome 10, analysis 1]

13. Secondary Outcome: Percentage of Participants Responding to Hepatitis B Surface Antigen
Description: Participant serum samples were collected for testing with an enhanced chemiluminescence assay for antibodies to Hepatitis B Surface Antigen. Response was defined as a titer >=10 mIU/mL.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 588 | 599 | 580 | 286 | 1767
Percentage of participants | 99.66 [98.78 to 99.96] | 100.00 [99.39 to 100.00] | 100.00 [99.37 to 100.00] | 98.95 [96.97 to 99.78] | 99.89 [99.59 to 99.99]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = -0.34, 95% CI 2-sided [-1.23 to 0.30] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = -0.34, 95% CI 2-sided [-1.23 to 0.32] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = 0.00, 95% CI 2-sided [-0.64 to 0.66] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 0.92, 95% CI 2-sided [0.20 to 2.90]

14. Secondary Outcome: Percentage of Participants Responding to Diphtheria Toxin
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to diphtheria toxin. Response was defined as a titer >=0.1 IU/mL.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 622 | 625 | 618 | 301 | 1865
Percentage of participants | 85.05 [82.00 to 87.76] | 84.80 [81.74 to 87.52] | 86.41 [83.45 to 89.01] | 87.71 [83.46 to 91.20] | 85.42 [83.73 to 86.99]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = 0.25, 95% CI 2-sided [-3.74 to 4.24] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = -1.35, 95% CI 2-sided [-5.26 to 2.57] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = -1.64, 95% CI 2-sided [-5.56 to 2.28] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = -2.35, 95% CI 2-sided [-6.02 to 2.09]

15. Secondary Outcome: Percentage of Participants Responding to Tetanus Toxin
Description: Participant serum samples were collected for testing with an ELISA for anti-tetanus antibodies. Response was defined as a titer >=0.1 IU/mL.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 622 | 609 | 612 | 300 | 1843
Percentage of participants | 99.84 [99.11 to 100.00] | 100.00 [99.40 to 100.00] | 100.00 [99.40 to 100.00] | 98.67 [96.62 to 99.64] | 99.95 [99.70 to 100.00]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot B) = -0.16, 95% CI 2-sided [-0.91 to 0.47] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot C) = -0.16, 95% CI 2-sided [-0.90 to 0.47] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot B - Lot C) = 0.00, 95% CI 2-sided [-0.63 to 0.62] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 1.28, 95% CI 2-sided [0.46 to 3.33]

16. Secondary Outcome: Percentage of Participants Responding to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. Response was defined as follows: 1) if the predose titer was <4 times the lower limit of quantitation (4X LLOQ) then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 596 | 585 | 580 | 289 | 1761
Percentage of participants | 99.33 [98.29 to 99.82] | 97.61 [96.02 to 98.69] | 98.97 [97.76 to 99.62] | 97.92 [95.54 to 99.23] | 98.64 [97.98 to 99.12]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = 1.73, 95% CI 2-sided [0.37 to 3.40] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = 0.36, 95% CI 2-sided [-0.77 to 1.63] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = -1.36, 95% CI 2-sided [-3.03 to 0.15] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 0.72, 95% CI 2-sided [-0.59 to 3.14]

17. Secondary Outcome: Percentage of Participants Responding to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 620 | 615 | 601 | 304 | 1836
Percentage of participants | 85.97 [82.98 to 88.61] | 87.32 [84.43 to 89.84] | 89.02 [86.24 to 91.40] | 92.11 [88.48 to 94.88] | 87.42 [85.81 to 88.90]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = -1.35, 95% CI 2-sided [-5.17 to 2.47] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = -3.06, 95% CI 2-sided [-6.79 to 0.67] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = -1.71, 95% CI 2-sided [-5.37 to 1.94] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = -4.70, 95% CI 2-sided [-7.73 to -0.86]

18. Secondary Outcome: Percentage of Participants Responding to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 590 | 574 | 560 | 286 | 1724
Percentage of participants | 81.19 [77.79 to 84.26] | 78.40 [74.80 to 81.70] | 78.75 [75.13 to 82.07] | 76.22 [70.86 to 81.04] | 79.47 [77.48 to 81.35]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = 2.77, 95% CI 2-sided [-1.83 to 7.39] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = 2.41, 95% CI 2-sided [-2.21 to 7.06] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = -0.36, 95% CI 2-sided [-5.14 to 4.42] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 3.28, 95% CI 2-sided [-1.70 to 8.85]

19. Secondary Outcome: Percentage of Participants Responding to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 613 | 611 | 594 | 298 | 1818
Percentage of participants | 86.95 [84.02 to 89.51] | 91.00 [88.44 to 93.15] | 91.08 [88.49 to 93.25] | 86.91 [82.55 to 90.53] | 89.66 [88.17 to 91.02]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot B) = -4.12, 95% CI 2-sided [-7.69 to -0.63] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot A - Lot C) = -4.17, 95% CI 2-sided [-7.75 to -0.66] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -10% and 10%; Response Rate Difference (Lot B - Lot C) = -0.07, 95% CI 2-sided [-3.32 to 3.20] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 2.85, 95% CI 2-sided [-0.85 to 7.36]

20. Secondary Outcome: Percentage of Participants Responding to Poliovirus Type 1
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 1. Response is defined as a titer >=8.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 630 | 632 | 628 | 307 | 1890
Percentage of participants | 100.00 [99.42 to 100.00] | 100.00 [99.42 to 100.00] | 100.00 [99.41 to 100.00] | 99.35 [97.67 to 99.92] | 100.00 [99.81 to 100.00]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot B) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot C) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot B - Lot C) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 0.66, 95% CI 2-sided [0.18 to 2.36]

21. Secondary Outcome: Percentage of Participants Responding to Poliovirus Type 2
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 2. Response is defined as a titer >=8.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 630 | 632 | 633 | 307 | 1895
Percentage of participants | 100.00 [99.42 to 100.00] | 100.00 [99.42 to 100.00] | 100.00 [99.42 to 100.00] | 100.00 [98.81 to 100.00] | 100.00 [99.81 to 100.00]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot B) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot C) = 0.00, 95% CI 2-sided [-0.61 to 0.60] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot B - Lot C) = 0.00, 95% CI 2-sided [-0.61 to 0.60] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 0.00, 95% CI 2-sided [-0.20 to 1.24]

22. Secondary Outcome: Percentage of Participants Responding to Poliovirus Type 3
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 3. Response is defined as a titer >=8.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lot A | V419 Lot B | V419 Lot C | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 624 | 625 | 625 | 304 | 1874
Percentage of participants | 100.00 [99.41 to 100.00] | 100.00 [99.41 to 100.00] | 100.00 [99.41 to 100.00] | 99.67 [98.18 to 99.99] | 100.00 [99.80 to 100.00]
Statistical Analysis 1: Comparison: V419 Lot A vs V419 Lot B; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot B) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 2: Comparison: V419 Lot A vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot A - Lot C) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 3: Comparison: V419 Lot B vs V419 Lot C; Test type: Non-Inferiority or Equivalence — Equivalence requires that the 2-sided 95% Confidence Intervals of the response rate difference are between -5% and 5%; Response Rate Difference (Lot B - Lot C) = 0.00, 95% CI 2-sided [-0.61 to 0.61] — Response rate difference was stratified by brand of birth dose of Hepatitis B vaccine
Statistical Analysis 4: Comparison: Control vs V419 Lots A, B, and C Combined; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 0.33, 95% CI 2-sided [0.05 to 1.85]

23. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had an infant vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 4.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1744 | 271 | 584 | 572 | 588
EU/mL | 110.61 [106.92 to 114.42] | 102.82 [93.70 to 112.82] | 110.41 [104.08 to 117.14] | 110.62 [104.14 to 117.51] | 110.79 [104.65 to 117.29]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, Analysis of Covariance; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.07, 95% CI 2-sided [0.98 to 1.17]

24. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1742 | 271 | 583 | 572 | 587
EU/mL | 106.30 [102.73 to 110.00] | 121.00 [110.19 to 132.87] | 101.81 [95.85 to 108.14] | 104.70 [98.66 to 111.12] | 112.60 [106.27 to 119.31]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.86, 95% CI 2-sided [0.79 to 0.95]

25. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1746 | 271 | 584 | 573 | 589
EU/mL | 104.51 [100.14 to 109.07] | 142.32 [126.68 to 159.89] | 94.26 [87.23 to 101.85] | 108.69 [101.41 to 116.51] | 111.42 [103.44 to 120.02]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p = 0.035, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.74, 95% CI 2-sided [0.66 to 0.83]

26. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 23
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1746 | 271 | 584 | 573 | 589
EU/mL | 451.04 [433.21 to 469.60] | 337.79 [299.43 to 381.05] | 409.37 [379.54 to 441.54] | 475.65 [444.85 to 508.59] | 471.52 [441.30 to 503.81]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.31, 95% CI 2-sided [1.17 to 1.46]

27. Secondary Outcome: Percentage of Participants Responding to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had a vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1616 | 254 | 535 | 531 | 550
Percentage of participants | 98.51 [97.80 to 99.05] | 98.43 [96.02 to 99.57] | 99.25 [98.10 to 99.80] | 98.12 [96.56 to 99.09] | 98.18 [96.68 to 99.12]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 0.12, 95% CI 2-sided [-1.11 to 2.58]

28. Secondary Outcome: Percentage of Participants Responding to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1669 | 261 | 559 | 550 | 560
Percentage of participants | 95.33 [94.20 to 96.29] | 95.40 [92.11 to 97.60] | 96.06 [94.10 to 97.52] | 94.36 [92.09 to 96.14] | 95.54 [93.48 to 97.09]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = -0.16, 95% CI 2-sided [-2.41 to 3.22]

29. Secondary Outcome: Percentage of Participants Responding to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1608 | 258 | 539 | 530 | 539
Percentage of participants | 92.16 [90.74 to 93.43] | 91.09 [86.92 to 94.26] | 91.28 [88.57 to 93.52] | 92.08 [89.44 to 94.23] | 93.14 [90.66 to 95.12]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 1.15, 95% CI 2-sided [-2.13 to 5.47]

30. Secondary Outcome: Percentage of Participants Responding to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1664 | 264 | 556 | 549 | 559
Percentage of participants | 92.97 [91.63 to 94.15] | 90.15 [85.90 to 93.47] | 91.91 [89.32 to 94.04] | 94.17 [91.87 to 95.98] | 92.84 [90.38 to 94.84]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (Comb - Ctrl) = 3.00, 95% CI 2-sided [-0.39 to 7.40]

31. Secondary Outcome: Geometric Mean Concentration of Antibodies to Pneumococcal Serotypes
Description: Participant serum samples were collected for testing with a multiplex electrochemiluminescence-based detection assay for serotype-specific pneumococcal polysaccharide antibodies. Analysis for this outcome included only non-inferiority of V419 Lots A, B, and C Combined versus Control.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V419 Lots A, B, and C Combined | Control | V419 Lot A | V419 Lot B | V419 Lot C
Number analyzed (Participants) | 1256 | 191 | 414 | 419 | 423
µg/mL
  Serotype 1 (n=1256, 191, 414, 419, 423) | 1.44 [1.38 to 1.50] | 1.55 [1.39 to 1.73] | 1.47 [1.36 to 1.59] | 1.40 [1.30 to 1.51] | 1.44 [1.34 to 1.55]
  Serotype 3 (n=1255, 191, 414, 418, 423) | 0.48 [0.46 to 0.50] | 0.50 [0.45 to 0.56] | 0.48 [0.45 to 0.51] | 0.48 [0.44 to 0.51] | 0.47 [0.44 to 0.50]
  Serotype 4 (n=1255, 189, 414, 418, 423) | 1.22 [1.17 to 1.27] | 1.22 [1.10 to 1.35] | 1.27 [1.18 to 1.36] | 1.16 [1.08 to 1.25] | 1.24 [1.16 to 1.34]
  Serotype 5 (n=1256, 191, 414, 419, 423) | 1.49 [1.42 to 1.57] | 1.61 [1.41 to 1.82] | 1.49 [1.36 to 1.64] | 1.49 [1.36 to 1.63] | 1.49 [1.36 to 1.63]
  Serotype 6A (n=1251, 191, 412, 417, 422) | 2.57 [2.45 to 2.69] | 2.96 [2.64 to 3.32] | 2.49 [2.29 to 2.71] | 2.66 [2.45 to 2.90] | 2.55 [2.36 to 2.75]
  Serotype 6B (n=1255, 190, 414, 419, 422) | 1.01 [0.94 to 1.09] | 1.29 [1.07 to 1.54] | 1.01 [0.88 to 1.14] | 1.01 [0.89 to 1.15] | 1.01 [0.89 to 1.14]
  Serotype 7F (n=1256, 191, 414, 419, 423) | 2.74 [2.64 to 2.85] | 3.08 [2.77 to 3.41] | 2.78 [2.60 to 2.97] | 2.75 [2.58 to 2.94] | 2.70 [2.53 to 2.87]
  Serotype 9V (n=1256, 189, 414, 419, 423) | 1.35 [1.29 to 1.41] | 1.35 [1.19 to 1.52] | 1.40 [1.29 to 1.52] | 1.30 [1.21 to 1.41] | 1.35 [1.25 to 1.46]
  Serotype 14 (n=1256, 191, 414, 419, 423) | 4.74 [4.48 to 5.01] | 4.83 [4.26 to 5.48] | 4.91 [4.45 to 5.42] | 4.85 [4.42 to 5.32] | 4.47 [4.05 to 4.93]
  Serotype 18C (n=1253, 191, 413, 418, 422) | 1.62 [1.55 to 1.69] | 1.82 [1.62 to 2.03] | 1.69 [1.57 to 1.82] | 1.62 [1.51 to 1.75] | 1.55 [1.44 to 1.67]
  Serotype 19A (n=1254, 191, 413, 418, 423) | 1.60 [1.53 to 1.68] | 1.75 [1.55 to 1.99] | 1.67 [1.55 to 1.81] | 1.52 [1.41 to 1.65] | 1.61 [1.49 to 1.74]
  Serotype 19F (n=1256, 191, 414, 419, 423) | 2.18 [2.10 to 2.27] | 2.26 [2.03 to 2.50] | 2.24 [2.09 to 2.41] | 2.11 [1.97 to 2.26] | 2.19 [2.05 to 2.33]
  Serotype 23F (n=1254, 190, 412, 419, 423) | 1.10 [1.04 to 1.16] | 1.20 [1.04 to 1.38] | 1.16 [1.05 to 1.28] | 1.07 [0.97 to 1.18] | 1.07 [0.97 to 1.19]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 1; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.92, 95% CI 2-sided [0.82 to 1.04]
Statistical Analysis 2: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 3; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.95, 95% CI 2-sided [0.84 to 1.06]
Statistical Analysis 3: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 4; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.00, 95% CI 2-sided [0.89 to 1.12]
Statistical Analysis 4: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 5; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.93, 95% CI 2-sided [0.80 to 1.07]
Statistical Analysis 5: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 6A; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.87, 95% CI 2-sided [0.77 to 0.99]
Statistical Analysis 6: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 6B; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p = 0.055, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.79, 95% CI 2-sided [0.64 to 0.96]
Statistical Analysis 7: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 7F; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.89, 95% CI 2-sided [0.80 to 0.99]
Statistical Analysis 8: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 9V; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 1.00, 95% CI 2-sided [0.88 to 1.13]
Statistical Analysis 9: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 14; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.95, 95% CI 2-sided [0.82 to 1.10]
Statistical Analysis 10: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 18C; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.89, 95% CI 2-sided [0.79 to 1.00]
Statistical Analysis 11: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 19A; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.91, 95% CI 2-sided [0.80 to 1.03]
Statistical Analysis 12: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 19F; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.97, 95% CI 2-sided [0.87 to 1.08]
Statistical Analysis 13: Comparison: V419 Lots A, B, and C Combined vs Control; Pneumococcal Serotype 23F; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 4]; GMC Ratio (Combined/Control) = 0.90, 95% CI 2-sided [0.77 to 1.06]

32. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reactions
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3 Solicited injection site reaction: Pain, Cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling, >5 cm. Grade 3 Solicited systemic reactions: Fever (Pyrexia), >=39.5°C rectal; Vomiting, >=6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal, >3 hours; Drowsiness (Somnolence), Sleeping most of the time or difficult to wake up; Appetite lost, Refuses >=3 feeds or refuses most feeds; Irritability, Inconsolable.
Time Frame: Up to 5 days after any infant vaccination (up to 6 months)
Population: Participants included in these analyses were All Subjects as Treated population and were defined as all vaccinated participants with safety follow up. This outcome applied only to V419 Lots A, B, and C Combined and Control; therefore, data for the individual V419 lots are not reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Control | V419 Lots A, B, and C Combined
Number analyzed (Participants) | 397 | 2390
Percentage of participants
  Any injection-site erythema | 40.8 | 44.6
  Severe injection-site erythema | 0.8 | 0.3
  Any injection-site pain | 72.0 | 70.0
  Severe injection-site pain | 5.5 | 6.0
  Any injection-site swelling | 34.5 | 34.5
  Severe injection-site swelling | 0.5 | 0.5
  Any crying abnormal | 72.5 | 74.8
  Severe crying abnormal | 12.6 | 9.5
  Any decreased appetite | 47.4 | 48.5
  Severe decreased appetite | 1.3 | 1.4
  Any irritability | 79.8 | 80.7
  Severe irritability | 6.5 | 7.8
  Any pyrexia | 33.2 | 47.1
  Severe pyrexia | 1.3 | 1.4
  Any somnolence | 73.3 | 73.2
  Severe somnolence | 3.0 | 3.5
  Any vomiting | 24.9 | 26.7
  Severe vomiting | 1.5 | 0.8

33. Secondary Outcome: Percentage of Participants With Elevated Temperature by Severity
Description: Maximum temperature (all routes) was based on actual temperatures recorded with no adjustments to the measurement route. Maximum temperature (rectal) was required of all participants if the reading by another method was >=38.0°C.
Time Frame: Up to 5 days after any infant vaccination (up to 6 months)
Population: Participants included in this analyses were All Subjects as Treated population defined as all vaccinated participants with safety follow up and temperature data. This outcome applied only to V419 Lots A, B, and C Combined and Control; therefore, data for the individual V419 lots are not reported.
Measure: Number; unit: Percentage of participants
Arm/Group | V419 Lots A, B, and C Combined | Control
Number analyzed (Participants) | 2308 | 378
Percentage of participants
  All routes <38.0°C | 50.8 [1.38 to 1.50] | 64.6 [1.39 to 1.73]
  All routes >=38.0°C and <38.5°C, mild | 27.2 [0.46 to 0.50] | 23.3 [0.45 to 0.56]
  All routes >=38.5°C and <39.5°C, moderate | 19.5 [1.17 to 1.27] | 10.8 [1.10 to 1.35]
  All routes >=39.5°C, severe | 2.4 [1.42 to 1.57] | 1.3 [1.41 to 1.82]
  Rectal <38.0°C | 47.7 [2.45 to 2.69] | 59.0 [2.64 to 3.32]
  Rectal >=38.0°C and <38.5°C, mild | 26.5 [0.94 to 1.09] | 23.0 [1.07 to 1.54]
  Rectal >=38.5°C and <39.5°C, moderate | 19.0 [2.64 to 2.85] | 10.6 [2.77 to 3.41]
  Rectal >=39.5°C, severe | 2.4 [1.29 to 1.41] | 1.3 [1.19 to 1.52]
Statistical Analysis 1: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference, all routes <38.0°C; Test type: Superiority or Other; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-18.8 to -8.4] — Mean Difference is V419 - Control. The 95% confidence interval is based on the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference, all routes >=38°C and <38.5°; Test type: Superiority or Other; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-0.9 to 8.3] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference, all routes >=38.5°C and <39.5°; Test type: Superiority or Other; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [4.8 to 11.9] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 4: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference, all routes >=39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.7 to 2.2] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 5: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference; rectal <38.0°C; Test type: Superiority or Other; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-16.6 to -5.9] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 6: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference; rectal >=38.0°C and <38.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-1.4 to 7.8] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 7: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference, rectal >=38.5°C and <39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [4.6 to 11.6] — [estimate comment as in outcome 33, analysis 1]
Statistical Analysis 8: Comparison: V419 Lots A, B, and C Combined vs Control; Estimated Difference, rectal >=39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.7 to 2.1] — [estimate comment as in outcome 33, analysis 1]

ADVERSE EVENTS:
Time Frame: SAEs: up to 6 months after vaccination 3 (the last infant vaccination) and up to 15 days after vaccination 4 (the toddler vaccination); Vaccine-related SAEs and deaths: up to Month 16 (duration of the study); Other AEs: up to 15 days after any vaccination
Description: The All Subjects as Treated population included all randomized participants who received at least one dose of study vaccine and had safety follow-up. For safety analysis, participants who received the 3 V419 lots were combined.
Arm/Group | V419 Lots A, B, and C Combined | Control
Serious Adverse Events (participants affected / at risk) | 94/2390 | 15/397
Other Adverse Events (participants affected / at risk) | 2259/2390 | 371/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V419 Lots A, B, and C Combined (N=2390) | Control (N=397)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Sudden infant death syndrome (General disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 9 (9) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 3 (3) | 0 (0)
Eczema herpeticum (Infections and infestations) | 1 (1) | 0 (0)
Gatroenteritis viral (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 12 (12) | 4 (4)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 4 (4) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V419 Lots A, B, and C Combined (N=2390) | Control (N=397)
Diarrhoea (Gastrointestinal disorders) | 192 (215) | 23 (24)
Vomiting (Gastrointestinal disorders) | 723 (1139) | 110 (171)
Crying (General disorders) | 1867 (4597) | 300 (763)
Irritability (General disorders) | 1993 (5595) | 324 (925)
Pyrexia (General disorders) | 1285 (2302) | 174 (274)
Otitis media (Infections and infestations) | 147 (162) | 39 (44)
Upper respiratory tract infection (Infections and infestations) | 276 (306) | 48 (54)
Decreased appetite (Metabolism and nutrition disorders) | 1355 (2586) | 217 (402)
Somnolence (Nervous system disorders) | 1816 (4497) | 298 (717)
Injection-site bruising (General disorders) | 128 (174) | 22 (31)
Injection-site erythema (General disorders) | 1302 (5189) | 203 (911)
Injection-site pain (General disorders) | 1883 (8854) | 314 (1815)
Injection-site swelling (General disorders) | 1073 (3652) | 166 (687)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.